CLINICAL TRIAL: NCT00235677
Title: A Blinded, Randomized, Sham-Controlled Trial of Endoscopic Gastroplication for the Treatment of Gastroesophageal Reflux Disease
Brief Title: Treatment Of Gastroesophageal Reflux Disease By Endoscopic Fundoplication, A Placebo-Controlled Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Endoplac
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Last update posted 2005-10-10 (Estimated); Status verified 2005-07

CONDITIONS: Gastroesophageal Reflux
Keywords: Endoscopic antireflux treatment; GERD; Sham-controlled; Endocinch
MeSH Terms: conditions — Gastroesophageal Reflux

INTERVENTIONS:
Procedure: Endoscopic gastroplication

SUMMARY:
Aim:

To evaluate the therapeutic efficacy of a therapeutic procedure, involving endoscopic suturing, for gastroesophageal reflux disease (GERD) compared to a sham procedure.

The hypotheses tested in this study were that active treatment would: 1) decrease the use of antisecretory medication, 2) decrease GERD symptoms, 3) improve quality of life, and 4) reduce esophageal acid exposure.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease (GERD) and the chronic, often lifelong, use of antisecretory medication have great clinical and economical implications for the patient, practicing physician and society in general. The currently available medication in GERD is very effective against heartburn, but less against the symptom of regurgitation. Surgical antireflux treatment offers a good alternative. The current surgical approach, a laparoscopic fundoplication, is safe and effective (a 90% reduction in use of antireflux medication), but in a significant subgroup of patients new symptoms arise (dysphagia, bloating) and perioperative morbidity, as well as financial costs are relatively high.

An endoscopic suturing system has been developed, offering a minimally invasive antireflux treatment, which can be performed in an outpatient setting. The procedure aims to create an endoscopic fundoplication, and could possibly serve as an alternative to antireflux medication and surgery. Recent, uncontrolled studies, have shown that the results of the endoscopic suturing system are satisfactory and that the procedure is safe.

This single-center, double-blinded, randomized, sham-controlled trial was conducted to evaluate the efficacy of endoscopic gastroplication by the Endocinch suturing system. Sixty patients with daily symptoms of GERD and abnormal esophageal 24-hr pH monitoring were randomly assigned to three endoscopic gastroplications (n = 20), to a sham procedure (n = 20) or to observation (n = 20). Primary endpoints were proton pump inhibitor use and GERD symptoms. Secondary endpoints were quality of life, 24-hr esophageal acid exposure, esophageal manometry and the occurrence of adverse events. Follow-up assessments were performed at 3 months. The research nurse and patients in the active and sham groups were blinded to the procedure assignment.

ELIGIBILITY:
Inclusion Criteria:

* typical symptoms of GERD (i.e., heartburn, regurgitation) for > 6 months,
* pathological esophageal acid exposure after discontinuation of medical therapy, proven by ambulatory 24-hour pH-monitoring with > 5% of time a pH < 4 and a symptom-association probability > 95% (19)
* patients considered for non-medical therapy, i.e. unwillingness to take life-long medication in medically-responding disease, suffering from medication side-effects or medically-intractable disease and unwillingness to undergo surgery
* willingness to accept a pre-treatment observation period of three months duration
* written informed consent

Exclusion Criteria:

* severe preexisting esophageal motility disorder (i.e., more than >40% non-transmitted or simultaneous contractions during a short esophageal manometry study)
* hiatal hernia (> 3 cm in length)
* history of antireflux or esophageal/gastric surgery
* severe psychiatric disease
* reflux esophagitis grade D (LA classification)
* Barrett's esophagus with dysplasia
* esophageal stenosis/malignancy
* pregnancy or lactation
* history of low therapeutic compliance
* other severe comorbidity (including cardiopulmonary disease, portal hypertension, collagen diseases, morbid obesity, coagulation disorder)
* use of anticoagulant or immunosuppressive drugs
* history of alcohol or drug abuse

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2003-08; Study Completion 2005-08

PRIMARY OUTCOMES:
Antisecretory drugs use
GERD symptoms (heartburn and regurgitation)

SECONDARY OUTCOMES:
Quality of life
24-hr esophageal acid exposure
Esophageal manometry
Occurrence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Matthijs P Schwartz, PhD, MD, Principal Investigator — UMC Utrecht; Andre J Smout, PhD, MD, Study Director — UMC Utrecht
Locations (1):
- Dept. of Gastroenterology, UMC Utrecht, Utrecht, Netherlands

REFERENCES:
- [Background] Schiefke I, Neumann S, Zabel-Langhennig A, Moessner J, Caca K. Use of an endoscopic suturing device (the "ESD") to treat patients with gastroesophageal reflux disease, after unsuccessful EndoCinch endoluminal gastroplication: another failure. Endoscopy. 2005 Aug;37(8):700-5. doi: 10.1055/s-2005-870128. PMID 16032486
- [Background] Arts J, Lerut T, Rutgeerts P, Sifrim D, Janssens J, Tack J. A one-year follow-up study of endoluminal gastroplication (Endocinch) in GERD patients refractory to proton pump inhibitor therapy. Dig Dis Sci. 2005 Feb;50(2):351-6. doi: 10.1007/s10620-005-1610-4. PMID 15745100
- [Background] Mahmood Z, McMahon BP, Arfin Q, Byrne PJ, Reynolds JV, Murphy EM, Weir DG. Endocinch therapy for gastro-oesophageal reflux disease: a one year prospective follow up. Gut. 2003 Jan;52(1):34-9. doi: 10.1136/gut.52.1.34. PMID 12477756
- [Background] Swain P, Park PO, Mills T. Bard EndoCinch: the device, the technique, and pre-clinical studies. Gastrointest Endosc Clin N Am. 2003 Jan;13(1):75-88. doi: 10.1016/s1052-5157(02)00106-x. PMID 12797428